CLINICAL TRIAL: NCT03887754
Title: Therapeutic Issues for Autism Spectrum Disorders: a Clinical Trial
Brief Title: Therapeutic Issues for Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Asmaa Salah, principal investigator, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Autism Spectrum Disorder
Record Dates: First submitted 2019-03-19; First posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Childhood Autism Rating Scale; Hyperbaric oxygen; Risperidone
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Risperidone; Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: Children were divided into four groups.Twenty autistic children in each group. They followed up for 2 years.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- The Hyperbaric oxygen therapy group (Active Comparator): This group consists of twenty autistic children received forty sessions of HBOT, the time of the session is one hour. The sessions were done at pressure 1.5 ATA (atmosphere absolute) and with 100% oxygen concentration, either in multiplace or monoplace chamber. The number of sessions per week allowed is five sessions per week, all participants were required to complete forty sessions within two months. After six months from the last session, another forty sessions would be taken in the same manner
  Interventions: Device: hyperbaric oxygen therapy
- The Risperidone group (Active Comparator): This group consists of twenty autistic children received Risperidone (dose: 0.25 mg per day in children weighing less than (20 kg); 0.5 mg per day in persons weighing more) for eight months.
  The medication schedule in the initial 2 months was based on the child's weight and clinical response. Adjusting the total daily dose according to response and/or adverse effects, at the end of these eight months of treatment we began the discontinuation phase. In this phase, gradual placebo substitution occurs. The discontinuation reduced the maintenance dose by 25% per week. Thus, the dose was 75% of the last week in the eight months for the first week, followed by 50% of the last week for the second week, 25% of the last week for the third week, and placebo only by the fourth week.
  Interventions: Drug: Risperidone
- The HBOT and Risperidone group (Active Comparator): This group consists of twenty autistic children received HBOT as the HBOT group in addition to Risperidone as the Risperidone group in the same manner and duration
  Interventions: Drug: Risperidone; Device: hyperbaric oxygen therapy
- The Control group (Placebo Comparator): This group consists of twenty autistic children received placebo in the form of multivitamins
  Interventions: Drug: Non specific Multivitamin

INTERVENTIONS:
Drug: Risperidone — It is antipsychotic drug used by dose: 0.25 mg per day in children weighing less than (20 kg); 0.5 mg per day in persons weighing more for 8 months.
  Other Names: Resperidal
  Arms: The HBOT and Risperidone group; The Risperidone group
Device: hyperbaric oxygen therapy — Sessions were done at pressure 1.5 ATA (atmosphere absolute) with 100% oxygen concentration, each lasting for one hour either in multiplace chamber or in monoplace chamber.
  Arms: The HBOT and Risperidone group; The Hyperbaric oxygen therapy group
Drug: Non specific Multivitamin — control group received non specific multivitamins as placebo for 8 months.
  Arms: The Control group

SUMMARY:
This study aimed to show the effects of hyperbaric oxygen therapy and/or Risperidone in improving symptoms of autism

DETAILED DESCRIPTION:
Autism spectrum disorders (ASDs) are clinical disorders with multiple developmental disabilities in skills associated with overall behavior and communication. The term (ASD) includes Autistic Disorder (AD), Pervasive Developmental Disorder-Not Otherwise Specified (PDD-NOS), and Asperger's Disorder .

Hyperbaric oxygen therapy (HBOT) is a treatment in which patients inside a hyperbaric chamber breathe a concentrated oxygen pressurized more than sea level (1 atmosphere absolute) .

It was obvious that autistic children may have some benefits of HBOT by increasing in cerebral perfusion during treatment. Inhalation of more pressurized oxygen might elevate partial pressure of oxygen in the arterial blood, and increased oxygen that reaches the brain . Another mechanism of action of HBOT that it might have anti-inflammatory properties by reduction of pro-inflammatory cytokines, interleukins 1 and 6, interferon-γ, and tumor necrosis factor-α. Furthermore, HBOT might enhance mitochondrial dysfunction, and upregulate the antioxidant enzymes production.

Risperidone is a second generation antipsychotic, approved by the Food and Drug Administration (FDA) for treatment of autism-related irritability. Its approved in 2006 only for children not less than 5 years old . This trial aimed to study the effects of hyperbaric oxygen therapy and/or Risperidone in management symptoms of autism.

ELIGIBILITY:
Inclusion Criteria:

* age of 5-7 years
* weight of at least 15 kg

Exclusion Criteria:

* Absence of significant medical problems and any other neuropsychiatric disorder requiring drug therapy (e.g., Bipolar disorder, psychosis).
* No concomitant treatment with psychotropic medication was allowed during the study.
* Weight less than 15 kg.
* Other cardiac, liver, gastrointestinal, renal, endocrine, blood and metabolic diseases

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Childhood Autism Rating Scale version 2 (CARS2)measured after one year and after two years to compare the effect of hyperbaric oxygen therapy, Risperidone, both of them and the placebo effect | two years
  The CARS is a 15 items behavioral rating scale developed to identify autism as well as to quantitatively describe the severity of the disorder. The items are as follows: I. Relating to People; II. Imitation; III. Emotional Response; IV. Body Use; V. Object Use; VI. Adaptation to Change; VII. Visual Response; VIII. Listening Response; IX. Taste; Smell, and Touch Response and Use; X. Fear or Nervousness; XI. Verbal Communication; XII. Nonverbal Communication; XIII. Activity Level; XIV. Level and Consistency of Intellectual Response; and XV. General Impressions. Each item is scored from 1 (no pathology) to 4 (severe pathology) in 0.5 intervals. A total score of 15-29.5 is considered non-autistic to minimal; a score of 30-36.5 is considered mild to moderate autism; a score of 37-60 is considered severe autism (these are based on raw scores)

CONTACTS AND LOCATIONS:
Overall Officials: Usama Aly, PhD, Study Chair — Minia University; Khaled Khaled, Prof., Study Director — Minia University

REFERENCES:
- [Background] Zulauf Logoz M. [The Revision and 5th Edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5): Consequences for the Diagnostic Work with Children and Adolescents]. Prax Kinderpsychol Kinderpsychiatr. 2014;63(7):562-76. doi: 10.13109/prkk.2014.63.7.562. German. PMID 25478714
- [Background] Lam G, Fontaine R, Ross FL, Chiu ES. Hyperbaric Oxygen Therapy: Exploring the Clinical Evidence. Adv Skin Wound Care. 2017 Apr;30(4):181-190. doi: 10.1097/01.ASW.0000513089.75457.22. PMID 28301358
- [Background] Calvert JW, Cahill J, Zhang JH. Hyperbaric oxygen and cerebral physiology. Neurol Res. 2007 Mar;29(2):132-41. doi: 10.1179/016164107X174156. PMID 17439697
- [Background] Rossignol DA, Bradstreet JJ, Van Dyke K, Schneider C, Freedenfeld SH, O'Hara N, Cave S, Buckley JA, Mumper EA, Frye RE. Hyperbaric oxygen treatment in autism spectrum disorders. Med Gas Res. 2012 Jun 15;2(1):16. doi: 10.1186/2045-9912-2-16. PMID 22703610
- [Background] LeClerc S, Easley D. Pharmacological therapies for autism spectrum disorder: a review. P T. 2015 Jun;40(6):389-97. PMID 26045648
- [Background] Starkstein SE, Vazquez S, Vrancic D, Nanclares V, Manes F, Piven J, Plebst C. SPECT findings in mentally retarded autistic individuals. J Neuropsychiatry Clin Neurosci. 2000 Summer;12(3):370-5. doi: 10.1176/jnp.12.3.370. PMID 10956571
- [Background] Bent S, Bertoglio K, Ashwood P, Nemeth E, Hendren RL. Brief report: Hyperbaric oxygen therapy (HBOT) in children with autism spectrum disorder: a clinical trial. J Autism Dev Disord. 2012 Jun;42(6):1127-32. doi: 10.1007/s10803-011-1337-3. PMID 21818676